CLINICAL TRIAL: NCT05650164
Title: A Multicenter, NI, Retrospective, Observational Study Evaluating Real-World Treatment Outcomes in Japanese Patients With Metastatic Renal Cell Carcinoma (mRCC) Treated With Avelumab Plus Axitinib as First-line Therapy: J-DART2
Brief Title: Treatment Outcomes in Japanese RCC Patients Treated With Avelumab Plus Axitinib as First-line Therapy: Retrospective Study (J-DART2)
Status: Completed | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991052; J-DART2 (Other: Alias Study Number)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Retrospective; Multicenter; Non-interventional; Medical chart review; Japan; Metastatic renal cell cancer(mRCC); Avelumab; Axitinib; First-line therapy; Standard care in real-world clinical setting
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — avelumab; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with metastatic renal cell carcinoma: Participants with metastatic renal cell carcinoma
  Interventions: Drug: avelumab; Drug: axitinib

INTERVENTIONS:
Drug: avelumab — as provided in real world practice
Drug: axitinib — as provided in real world practice

SUMMARY:
This study is a multicenter, non-interventional, retrospective, medical chart review of participants with metastatic renal cell cancer(mRCC) treated with avelumab plus axitinib as a first-line therapy in Japan between 20 December 2019 and 17 October 2022. All decisions regarding clinical management and treatment of the participating patients were made by the investigator as part of standard care in real-world clinical setting and were not contingent upon the patient's participation in the study. Data will be collected if available per study site.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoses of mRCC based on the General Rule for Clinical and Pathological Studies on RCC (Fifth Edition) before receiving avelumab plus axitinib as first-line therapy. Patients with mRCC who have unresectable disease, either unresectable locally advanced or metastatic disease.
2. Age over 18 years at the time of the first administration of avelumab plus axitinib as firstline therapy for mRCC (baseline).
3. Index date from 20 December 2019 to 17 October 2022.

Exclusion Criteria:

1. Patients participating in a prospective interventional clinical trial assessing an investigational product during the observation period.
2. Patients (or a patient's legally representative) refusing to provide patient data during the consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic renal cell cancer(mRCC) treated with avelumab plus axitinib as a first-line therapy in Japan between 20 December 2019 and 17 October 2022
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (19):
- Japan (19):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kochi Medical School Hospital, Nankoku, Kochi
  - National Hospital Organization Kyoto Medical Center, Kyoto, Kyoto
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Jichi Medical University Saitama Medical Center, Saitama, Saitama
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamagata University Hospital, Yamagata, Yamagata
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=B9991052
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Metastatic Renal Cell Carcinoma: Participants with metastatic renal cell carcinoma who were treated using avelumab plus axitinib as a first-line therapy.
Period: Overall Study
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Started | 171
Completed | 171
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 112
  >=65 years | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 170

OUTCOME MEASURES:

1. Primary Outcome: Age of Participants at Baseline
Description: The age of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: years
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
years | 71.0 [33 to 87]

2. Primary Outcome: Height of Participants at Baseline
Description: The height of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria. Here, number analyzed represents the number of participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 169
centimeters | 163.23 (8.60)

3. Primary Outcome: Body Weight of Participants at Baseline
Description: The body weight of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 169
kilograms | 63.117 (12.642)

4. Primary Outcome: Body Mass Index of Participants at Baseline
Description: The body mass index (BMI) of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram per square meter
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 169
kilogram per square meter | 23.593 (3.798)

5. Primary Outcome: C-Reactive Protein Levels of Participants at Baseline
Description: The C-reactive protein levels of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 167
milligrams per liter | 1.575 (3.001)

6. Primary Outcome: Estimated Glomerular Filtration Rate of Participants at Baseline
Description: The estimated Glomerular Filtration Rate (eGFR) is an index of kidney function. eGFR was calculated using factors such as serum creatinine level, age, sex, and in millimeter per minute per 1.73 square meter (ml/min/1.73 m^2), and tabulated in three categories (<60, ≥60, unknown). An eGFR <60 indicates some degree of kidney impairment. And eGFR > 60 is generally considered to be within the normal range.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  Less than 60 | 124
  More than or equal to 60 | 45
  Unknown | 1

7. Primary Outcome: Smoking History Status of Participants at Baseline
Description: The smoking history status of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No (no past smoking) | 67
  No (history of past smoking) | 62
  Yes | 26
  Unknown | 15

8. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Scale Score Status of Participants at Baseline
Description: ECOG-PS assessed participant's performance status on a 5 point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2= ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 169
Participants
  0 | 132
  1 | 25
  2 | 5
  3 | 6
  4 | 1

9. Primary Outcome: Number of Participants With Metastatic Organs at Baseline
Description: The Number of participants with Metastatic Organs of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  Lung | 101
  Liver | 13
  Bone | 28
  Brain | 3
  Regional lymph node | 22
  Distant lymph node | 19
  Other | 45

10. Primary Outcome: Invasion Depth (T Factor) of Participants at Baseline
Description: TX: Primary tumor cannot be assessed, T0: No evidence of primary tumor, T1: Tumor ≤7 cm in greatest dimension, limited to the kidney, T1a: Tumor≤4cm in greatest dimension, limited to the kidney, T1b: Tumor>4 cm but ≤7 cm in greatest dimension, limited to the kidney, T2: Tumor >7 cm in greatest dimension, limited to the kidney, T2a: Tumor >7 cm but ≤10 cm in greatest dimension, limited to the kidney, T2b: Tumor >10 cm, limited to the kidney, T3: Tumor extends into major veins or perinephric tissues, but not into the ipsilateral adrenal gland and not beyond Gerota's fascia,T3a: Tumor extends into the renal vein or its segmental branches, or invades the pelvicalyceal system, or invades perirenal and, T3b: Tumor extends into the vena cava below the diaphragm, T3c: Tumor extends into the vena cava above the diaphragm or invades the wall of the vena cava, T4: Tumor invades beyond Gerota's fascia (including contiguous extension into the ipsilateral adrenal gland)
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Efficacy Analysis Set is a subset of the FAS comprising patients whose index date is prior to April 30, 2022, to ensure a 6-month follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 150
Participants
  TX | 6
  T0 | 0
  T1 | 1
  T1a | 26
  T1b | 29
  T2 | 2
  T2a | 6
  T2b | 2
  T3 | 2
  T3a | 43
  T3b | 10
  T3c | 2
  T4 | 10
  Unknown | 11

11. Primary Outcome: Lymph Node Metastasis (N Factor) Status of Participants at Baseline
Description: Lymph node metastasis (N factor) of participants at baseline was reported. NX: Regional lymph nodes cannot be assessed, N0: No regional lymph node metastasis, N1: Metastasis in regional lymph node(s).
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  NX | 7
  N0 | 127
  N1 | 30
  Unknown | 6

12. Primary Outcome: Distant Metastasis (M Factor) Status of Participants at Baseline
Description: Distant metastasis (M factor) of participants at baseline was reported. M0: No distant metastasis, M1: Distant metastasis.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  MX | 0
  M0 | 20
  M1 | 150
  Unknown | 0

13. Primary Outcome: Tumor Histological Type of Participants at Baseline
Description: Tumor histological type of participants at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  Clear cell renal cell carcinoma | 154
  Papillary renal cell carcinoma | 4
  Chromophobe renal cell carcinoma | 2
  Other | 4
  Unknown | 6

14. Primary Outcome: Number of Participants With Presence or Absence of Sarcomatoid Component in Participants at Baseline
Description: Number of Participants with Presence or Absence of Sarcomatoid Component at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria. . Here "Number of Participants Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 169
Participants
  Presence | 11
  Absence | 158

15. Primary Outcome: Fuhrman Grade Status of Participants at Baseline
Description: The four-tiered Fuhrman grading evaluates nuclear size, nuclear shape and presence of nucleolar prominence. Grade 1: small (=10 micrometer [mcm]) nuclear diameter, round/uniform nuclear shape and absent/inconspicuous nucleoli; Grade 2: large (=15 mcm) nuclear diameter, irregular outline nuclear shape and visible at *400 magnification nucleoli; Grade 3: larger (=20 mcm) nuclear diameter, obvious irregular outline nuclear shape and visible and prominent at *100 magnification nucleoli; Grade 4: grade 3 plus bizarre multilobed nuclei +/- spindle cells. Participants whose Fuhrman Grade were not known were reported against "Unknown'.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  Grade 1 | 57
  Grade 2 | 0
  Grade 3 | 33
  Grade 4 | 16
  Unknown | 64

16. Primary Outcome: Availability of Proteinuria in Participants at Baseline
Description: Proteinuria is the presence of an excess of serum proteins in the urine, which may be an early sign of kidney disease. Here, negative (-)= <15 milligrams per deciliter (mg/dL) (Normal), positive (±) =15-29 mg/dL (increased risk for kidney disease), (1+) = 30 mg/dL(Early stages of kidney disease), (2+)= 100 mg/dL (Underlying kidney disease), (3+)= 300 mg/dL (kidney dysfunction).
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  minus (-) | 92
  plus minus (+-) | 22
  1+ | 17
  2+ | 6
  3+ | 6
  Not measured | 27

17. Primary Outcome: Performance of Nephrectomy in Participants
Description: Performance of nephrectomy at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 45
  Yes | 125
  Unknown | 0

18. Primary Outcome: Number of Participants With Presence or Absence of Clinically Important Comorbidities of Participants at Baseline
Description: Number of Participants with Presence or absence of clinically important comorbidities at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 59
  Yes | 111
  Unknown | 0

19. Primary Outcome: Number of Participants With Presence or Absence of Clinically Important Concomitant Drugs in Participants at Baseline
Description: Number of participants with Presence or absence of clinically important concomitant drugs at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 75
  Yes | 95
  Unknown | 0

20. Primary Outcome: Number of Participants With Initiation of Systemic Therapy Within One Year of Diagnosis
Description: Number of Participants with Initiation of Systemic Therapy within One Year of Diagnosis was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 81
  Yes | 89

21. Primary Outcome: Number of Participants With Karnofsky Performance Status Less Than (<) 80 Percent (%) at Baseline
Description: Karnofsky performance score was used to quantify participant's general well-being and activities of daily life and participants were classified based on their functional impairment. Karnofsky performance score ranges between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 157
  Yes | 13

22. Primary Outcome: Number of Participants With Hemoglobin Value Below the Lower Normal Limit at Baseline
Description: Number of participants with Hemoglobin value below the lower normal limit at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 85
  Yes | 85

23. Primary Outcome: Number of Participants With Corrected Calcium Value Above the Upper Normal Limit in Participants at Baseline
Description: Number of participants with Corrected calcium value above the upper normal limit at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 150
  Yes | 20

24. Primary Outcome: Number of Participants With Neutrophil Count Above the Upper Normal Limit in Participants at Baseline
Description: Number of Participants with Neutrophil count above the upper normal limit at baseline was reported.
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  No | 146
  Yes | 24

25. Primary Outcome: International Metastatic RCC Database Consortium (IMDC) Risk Group in Participants at Baseline
Description: IMDC criteria had 6 risk factors: Karnofsky Performance Status less than (<) 80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <1 year; corrected serum calcium; neutrophils and platelets more than (>) upper limit of normal (ULN); hemoglobin <lower limit of normal (LLN). Present risk factors were added, and then participants were stratified as: Low risk (0 factor), Medium risk (1-2 factors), High risk (more than or equal to [>=]3 factors).
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  Low risk | 44
  Medium risk | 92
  High risk | 34

26. Primary Outcome: Number of Risk Factors in Participants at Baseline
Description: Number of risk factors in participants at baseline was reported
Time Frame: At Baseline (prior to initial treatment with avelumab plus axitinib)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 170
Participants
  0 | 44
  1 | 50
  2 | 42
  3 | 21
  4 | 12
  5 | 1
  6 | 0

27. Secondary Outcome: Real-World Progression-Free Survival (Rw-PFS)
Description: rwPFS is defined as: The time from start of avelumab plus axitinib therapy to date of first disease progression (as clinically assessed by local investigator based on radiology, laboratory evidence, pathology, or other assessments) or death due to any cause, whichever occurred first.
Time Frame: From index date up to 31 Oct 2022, where index date was date of first prescription for avelumab plus axitinib between 20 December 2019 and 17 October 2022 (maximum observation period was of 34 months approximately)
Population: The efficacy analysis set is a subset of the FAS that includes patients whose index date is prior to 30 April 2022 to ensure a 6-months follow-up period.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 150
months | 13.8 [12.5 to 18]

28. Secondary Outcome: Time to Treatment Discontinuation (TTD)
Description: TTD is defined as the time from the start of treatment with avelumab plus axitinib to the end of treatment due to any cause except the effectiveness of the treatment.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 150
months | 17.2 [11.2 to 23.0]

29. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the start of treatment with avelumab plus axitinib to the date of death due to any cause. If there are no clinical records of death, the date when the patient was last documented to be alive will be confirmed based on medical records. The data will be censored at the date of last contact.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 150
months | 18.7 [16.3 to 20.6]

30. Secondary Outcome: Percentage of Participants With Best Overall Response of CR or PR (Objective Response Rate)
Description: The ORR is defined as the proportion of participants with a documented BOR (complete response (CR) or partial response (PR)) by the investigator during treatment with avelumab plus axitinib as firstline therapy. The BOR is defined as the best tumor response recorded during the observation period. The definitions of tumor responses are as follows: Complete or PR as the best adjudication result (CR > PR > stable disease [SD] > progressive disease [PD], not Evaluable [NE]) complies with the RECIST tumor assessment guidelines as closely as possible in clinical practice.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 150
percentage of participants | 53.3 [44.6 to 62.0]

31. Secondary Outcome: Number of Participants With Best Overall Response (BOR) for Primary Lesions
Description: BOR is the best tumor response recorded during observation period.Tumor response are defined as follows:Complete or PR as the best adjudication result (CR > PR > stable disease [SD] > progressive disease [PD],not Evaluable[NE]) in a method complied with RECIST version. 1.1tumor assessment as closely as possible in clinical practice by investigator's judgment.CR:Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR:Atleast 30% decrease in sum of diameters of target lesions,taking as reference the baseline sum diameters.SD:Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,taking as reference the smallest sum diameters. PD:atleast a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: as for outcome 27
Population: The efficacy analysis set is a subset of the FAS that includes patients whose index date is prior to 30 April 2022 to ensure a 6-months follow-up period. Here "Number of Participants Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
Number analyzed (Participants) | 135
Participants
  CR | 12
  PR | 60
  SD | 48
  PD | 14
  NE | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to approximately 34 months and 11 days. Serious and Other Adverse Events were not monitored/assessed in this study.
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Participants With Metastatic Renal Cell Carcinoma
All-Cause Mortality (participants affected / at risk) | 19/150
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT05650164/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT05650164/SAP_001.pdf